CLINICAL TRIAL: NCT00746629
Title: Behavioral Skill Adherence in Pediatric Obesity Treatment
Brief Title: Familial Overweight: Comparing Use of Strategies
Acronym: FOCUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seattle Children's Hospital (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Brian Saelens, Investigator, Seattle Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HD54871 (completed); 1R21DK095676 (NIH)
Record Dates: First submitted 2008-09-03; First posted 2008-09-04 (Estimated); Last update posted 2015-05-21 (Estimated); Status verified 2015-05

CONDITIONS: Overweight and Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prescribed Skills (Active Comparator): Behavioral skills are all prescribed and considered necessary tools expected to be used consistently, completely, and uniformly by all participants throughout treatment
  Interventions: Behavioral: FOCUS
- Self-Directed Skills (Experimental): Behavioral skills are considered a tool box from which families are encouraged to select skills that best apply to that family's situation in attempts to help their child make eating and activity change.
  Interventions: Behavioral: FOCUS

INTERVENTIONS:
Behavioral: FOCUS — Treatment will be delivered over a 20-week period. Participating children and at least one of their parents will attend weekly in-person clinic sessions. Treatment will consist of 20-25 minute meetings between the assigned interventionist and each child/parent pair to individualize treatment, with an emphasis on helping the family change eating and activity behaviors. Family meetings will be followed by separate child and parent group meetings lasting approximately 35-45 minutes. In both approaches, parents serve as primary implementers of the treatment for the child and, if overweight, for themselves. Group sessions provide education in diet and physical activity, parenting, and behavioral skills, although conditions differ in whether skills are "prescribed" or "self-directed". Children and parents will be weighed at each clinic visit.

SUMMARY:
The purpose of this study is to compare the efficacy of two different approaches (prescribed & self-directed) to the treatment of childhood obesity and their relative impact on child weight status, physical activity, and diet.

DETAILED DESCRIPTION:
Pediatric obesity is a highly prevalent problem, requiring both treatment and prevention efforts to reduce cardiovascular disease risk and metabolic consequences among affected children and the child population. The efficacy of family-based behavioral pediatric obesity treatment is likely compromised by non-optimal parent and child behavioral skills use (BSU). In pediatric obesity treatment trials, BSU assessment is infrequent, incomplete, and has unknown reliability. Poor and incomplete BSU measurement precludes improving behavioral interventions for pediatric obesity. Furthermore, different approaches to help families initiate and sustain BSU during and following treatment have not been tested. This study aims to investigate 1) prospective relations between BSU measured during and following treatment and change in child weight status, physical activity, and diet, and 2) differences in BSU trajectory between two different implementation approaches during and following treatment. Eighty-two parent-child (7-11 y.o.) pairs will participate in a 20-week treatment with follow-up at 3 and 6 months. Participants will be randomly assigned to receive either a prescriptive or self-directed implementation approach to family-based behavioral pediatric obesity treatment. BSU (monitoring, contingency management, environmental control) will be reported or assessed at pre-treatment, at the 5th, 10th, and 15th treatment sessions, at post-treatment and at the 3-month and 6-month follow-ups by the parent, interventionist, and supplemental evaluator. Prospective associations between BSU, measured multiple times and by multiple informant/formats, and change in child weight status (z-BMI) and weight-related behaviors (diet, physical activity) over the course of treatment and throughout follow up will be examined. This proposal will provide important information about the type of BSU and its measurement that is most related to short- and long-term treatment efficacy, and provide pilot data on the relative efficacy of different implementation approaches to initiate and sustain BSU in pediatric obesity intervention.

ELIGIBILITY:
Inclusion Criteria:

* Child age: 7-11 years.
* English-speaking.
* Parent is willing and able to actively participate in treatment.
* Overweight child: at or above 85th percentile for age- and gender-specific BMI, but not more than 175% above median BMI for age and gender.
* Overweight parent: BMI≥ 25.
* Live within 50 miles of Children's Hospital and Regional Medical Center.

Exclusion Criteria:

* Medical condition known to promote obesity (e.g. Prader-Willi syndrome, Cushing's syndrome).
* Already involved with another weight control program.
* Consistently engaging in weight-affecting behaviors (e.g. child: smoking)
* Significant diagnosed obesity-related co-morbidities (e.g. Type 2 diabetes)
* Taking weight-affecting medications (e.g. Ritalin)
* Participating parent or child: an existing thought disorder, suicidality, substance abuse disorder, or other psychological or medical conditions that may preclude full participation.
* Participating parent or child: Disability or illness that would preclude them from engaging in at least moderate intensity physical activity.
* Participating parent or child: Current or prior diagnosed eating disturbance.

Ages: 7 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 72 (Actual)
Dates: Start 2008-05; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Child weight status, physical activity, & diet. | 6 Months

SECONDARY OUTCOMES:
Secondary outcomes will include parents' BMI, and parents' physical activity and eating behaviors and covariates will include child age, gender, and household income. | 6 Months

CONTACTS AND LOCATIONS:
Overall Officials: Brian E Saelens, PhD, Principal Investigator — Seattle Children's Hospital
Locations (1):
- Seattle Children's Hospital Research Institute, Seattle, Washington, United States

REFERENCES:
- [Result] Saelens BE, Lozano P, Scholz K. A randomized clinical trial comparing delivery of behavioral pediatric obesity treatment using standard and enhanced motivational approaches. J Pediatr Psychol. 2013 Oct;38(9):954-64. doi: 10.1093/jpepsy/jst054. Epub 2013 Jul 31. PMID 23902797